CLINICAL TRIAL: NCT06345339
Title: A Phase 2/3 Multicenter, Double Blinded, Randomized, Dose-conversion, Active Control Study Examining the Efficacy and Safety of Armour Thyroid Compared to Synthetic T4 for the Treatment of Adults With Primary Hypothyroidism
Brief Title: A Study to Assess the Safety and Efficacy of Oral Armour Thyroid Compared to Synthetic T4 for the Treatment of Primary Hypothyroidism in Adult Participants
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-341
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Armour Thyroid; Synthetic T4
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Thyroid (USP); Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will receive Armour Thyroid for up to 81 weeks.
  Interventions: Drug: Armour Thyroid
- Group 2 (Experimental): Participants will alternate between Armour Thyroid and synthetic T4 for up to 81 weeks.
  Interventions: Drug: Armour Thyroid; Drug: Levothyroxine

INTERVENTIONS:
Drug: Armour Thyroid — Oral Capsule or Tablet
  Other Names: AGN-282176
Drug: Levothyroxine — Oral Capsule
  Other Names: Synthetic T4
  Arms: Group 2

SUMMARY:
This study will evaluate the efficacy and safety of Armour Thyroid treatment compared with synthetic T4 in subjects who have primary hypothyroidism and are currently stabilized (i.e., in-range thyroid-stimulating hormone [TSH]) on synthetic T4 treatment. This study will also therefore evaluate the efficacy and safety of dose conversion from synthetic T4 therapy to Armour Thyroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of primary hypothyroidism made >= 12 months prior to Screening.
* Be on continuous thyroid replacement therapy of synthetic T4 for primary hypothyroidism for at least 12 months immediately prior to the Screening Visit.
* Be on a stable FDA-approved daily dose of synthetic T4 prior to the Screening visit, and must be taking synthetic T4 dose of at least 25 mcg at Screening visit. Must enter the study using the same stable dose to determine dose conversion.
* Documentation of 1 in-range thyroid-stimulating hormone (TSH) (i.e., within 0.45 - 4.12 mIU/L, inclusive) at Screening and at least 1 additional in range TSH (i.e., within 0.45 - 4.12 mIU/L, inclusive) taken at a minimum of 6 weeks and a maximum of 12 months prior to Screening.

Exclusion Criteria:

* Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of Armour Thyroid or synthetic T4.
* History of alcohol or other substance abuse within the previous 6 months prior to the Screening.
* Known or suspected allergy or intolerance to any ingredients of Armour Thyroid, including its excipients, synthetic T4, other thyroid replacement medications, or pork products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Thyroid-Stimulating Hormone (TSH) Response | Week 55
  TSH response is defined as TSH values falling within 0.45 to 4.12 mIU/L (inclusive). TSH response will be determined at Week 55 and at a prior visit with no out-of-range TSH values in between (response rate is tested against a specified non-inferiority margin).
Number of Participants with Adverse Events (AEs) | Up to approximately 90 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve TSH Response | Week 55
  TSH response is defined as TSH values falling within 0.45 to 4.12 mIU/L. TSH response will be determined at Week 55 and at a prior visit with no out-of-range TSH values in between (response rate is tested against a specified non-inferiority margin [stricter than the one used in the Primary Outcome Measure]).
Number of Participants Needing Altered Dose Conversion from Synthetic T4 to Armour Thyroid | Up to approximately 29 weeks
  Number of participants needing altered dose conversion from synthetic T4 to Armour Thyroid.
Frequency of Dose Titrations During the Double-Blind (DB) Period Among Participants who Achieved TSH Response at the End of the DB Period | Week 55
  Frequency of dose titrations (0,1,2...) during the DB period among participants who achieved TSH response at the end of the DB period.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (139):
- United States (134):
  - Central Research Associates /ID# 255719, Birmingham, Alabama
  - UAB Hospital /ID# 262565, Birmingham, Alabama
  - Kaiser San Diego Dept Endocrinology, SCPMG /ID# 262552, Bonita, California
  - Facey Medical Foundation - Burbank /ID# 262104, Burbank, California
  - John Muir Medical Center /ID# 257103, Concord, California
  - Diagnamics Inc. /ID# 262680, Encinitas, California
  - Providence - St. Jude Medical Center /ID# 256520, Fullerton, California
  - NorCal Medical Research /ID# 256512, Greenbrae, California
  - Velocity Clinical Research - Huntington Park /ID# 259044, Huntington Park, California
  - Scripps Whittier Diabetes Institute /ID# 259215, La Jolla, California
  - Facey Medical Foundation /ID# 260863, Mission Hills, California
  - Hoag Memorial Hospital Presbyterian /ID# 260990, Newport Beach, California
  - Diabetes Associates Medical Group /ID# 256949, Orange, California
  - Western University of Health Sciences /ID# 262183, Pomona, California
  - Research at Mills-Peninsula Medical Center - Sutter Health /ID# 258825, San Mateo, California
  - Care Access - Santa Clarita /ID# 262573, Santa Clarita, California
  - Facey Medical Foundation - Valencia /ID# 262102, Santa Clarita, California
  - Olive View UCLA Medical Center /ID# 259092, Sylmar, California
  - The Lundquist Institute at Harbor-UCLA Medical Center /ID# 262572, Torrance, California
  - Diablo Clinical Research /ID# 261329, Walnut Creek, California
  - San Fernando Valley Health Institute /ID# 257363, West Hills, California
  - New England Research Associates - Bridgeport /ID# 262184, Bridgeport, Connecticut
  - Innovative Research of West Florida /ID# 257356, Clearwater, Florida
  - ALL Medical Research /ID# 256748, Cooper City, Florida
  - Northeast Research Institute (NERI) /ID# 261841, Fleming Island, Florida
  - Northeast Research Institute (NERI) /ID# 261846, Fleming Island, Florida
  - The Center for Diabetes and Endocrine Care /ID# 255721, Fort Lauderdale, Florida
  - Encore Medical Research LLC /ID# 256758, Hollywood, Florida
  - East Coast Institute For Research - LaVilla - West Monroe Street /ID# 256972, Jacksonville, Florida
  - The University of Florida Heal /ID# 257361, Jacksonville, Florida
  - East Coast Research - Jacksonville /ID# 256971, Jacksonville, Florida
  - Encore Research Group-Jacksonville Center for Clinical Research /ID# 256147, Jacksonville, Florida
  - Baptist Health Research Institute /ID# 260989, Jacksonville, Florida
  - South Florida Wellness & Clinic /ID# 256513, Margate, Florida
  - Med Research of Florida /ID# 257837, Miami, Florida
  - Ocean Blue Medical Research Center, Inc /ID# 260438, Miami Springs, Florida
  - Adult Medicine of Lake County - Mount Dora /ID# 257371, Mt. Dora, Florida
  - Suncoast Clinical Research Pasco County /ID# 257018, New Port Richey, Florida
  - West Orange Endocrinology /ID# 256139, Ocoee, Florida
  - Suncoast Clinical Research - Palm Harbor /ID# 256741, Palm Harbor, Florida
  - Comprehensive Medical & Research Center /ID# 261678, Plantation, Florida
  - Northeast Research Institute - St. Augustine /ID# 261857, Saint Augustine, Florida
  - Metabolic Research Inst /ID# 255729, West Palm Beach, Florida
  - Grady Clinical Research Center Grady Memorial Hospital /ID# 258419, Atlanta, Georgia
  - Atlanta Diabetes Associates /ID# 255736, Atlanta, Georgia
  - East Coast Institute for Research - Canton /ID# 256974, Canton, Georgia
  - Centricity Research - Endocrine Consultants Research /ID# 255738, Columbus, Georgia
  - Physicians Research Associates, LLC /ID# 255675, Lawrenceville, Georgia
  - The Jones Center Clinical Research /ID# 256529, Macon, Georgia
  - Endocrine Research Solutions /ID# 256784, Roswell, Georgia
  - Pacific Diabetes & Endocrine Center /ID# 259030, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, LLC /ID# 256753, Idaho Falls, Idaho
  - Northwestern University Feinberg School of Medicine /ID# 260677, Chicago, Illinois
  - West Broadway Clinic /ID# 256756, Council Bluffs, Iowa
  - Iowa Diabetes and Endocrinology Research Center /ID# 256750, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology /ID# 256749, Topeka, Kansas
  - University of Louisville Hospital /ID# 262568, Louisville, Kentucky
  - Robley Rex VA Medical Center /ID# 262569, Louisville, Kentucky
  - L-MARC Research Center /ID# 255733, Louisville, Kentucky
  - Pennington Biomedical Research Center /ID# 262390, Baton Rouge, Louisiana
  - Nola Care Clinical Research /ID# 260145, Metairie, Louisiana
  - Omega Clinical Research /ID# 260162, Metairie, Louisiana
  - Tufts Medical Center /ID# 262974, Boston, Massachusetts
  - Circle Health Diabetes and Endocrine Center /ID# 270461, Dracut, Massachusetts
  - NECCR PrimaCare Research, LLC /ID# 256531, Fall River, Massachusetts
  - Metro Detroit Endocrinology Center /ID# 260862, Dearborn, Michigan
  - Michigan Healthcare Professionals /ID# 260859, Farmington Hills, Michigan
  - Elite Clinical Research Center /ID# 256782, Flint, Michigan
  - Diabetes and Endocrinology Specialists /ID# 259068, Chesterfield, Missouri
  - University of Missouri Hospital /ID# 262562, Columbia, Missouri
  - Jefferson City Medical Group /ID# 257099, Jefferson City, Missouri
  - Mercy Research - Springfield /ID# 262385, Springfield, Missouri
  - St. Louis University /ID# 262375, St Louis, Missouri
  - Washington University-School of Medicine /ID# 262391, St Louis, Missouri
  - Billings Clinic /ID# 258316, Billings, Montana
  - Mercury Street Medical /ID# 259632, Butte, Montana
  - Bryan Health Pine Lake Campus /ID# 259638, Lincoln, Nebraska
  - Methodist Physicians Clinic /ID# 259276, Omaha, Nebraska
  - Palm Research Center /ID# 256131, Las Vegas, Nevada
  - Northern Nevada Endocrinology /ID# 259646, Reno, Nevada
  - Southern New Hampshire Diabetes and Endocrinology /ID# 257841, Nashua, New Hampshire
  - Albany Medical College- Endocrinology Washington Extension /ID# 256794, Albany, New York
  - Research Foundation of SUNY - University of Buffalo /ID# 261019, Buffalo, New York
  - NYC Research /ID# 258662, New York, New York
  - Endocrine Assc Long Island PC /ID# 257357, Smithtown, New York
  - Physician's East Endocrinology /ID# 256491, Greenville, North Carolina
  - Carteret Medical Group /ID# 256869, Morehead City, North Carolina
  - Lucas Research /ID# 256127, Morehead City, North Carolina
  - Lucas Research /ID# 257061, Morehead City, North Carolina
  - Accellacare - Salisbury /ID# 257019, Salisbury, North Carolina
  - Accellacare Wilmington /ID# 256744, Wilmington, North Carolina
  - Diabetes and Endocrinology Associates of Stark County Inc /ID# 256751, Canton, Ohio
  - Cleveland Clinic - Cleveland /ID# 262392, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - CarePoint East /ID# 264061, Columbus, Ohio
  - Lynn Institute of Norman /ID# 256785, Norman, Oklahoma
  - Lynn Institute of Oklahoma City /ID# 263141, Oklahoma City, Oklahoma
  - Diabetes & Endocrinology Consultants of Pennsylvania /ID# 259064, Feasterville-Trevose, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 256834, Philadelphia, Pennsylvania
  - Jefferson Health - Roosevelt Boulevard /ID# 256837, Philadelphia, Pennsylvania
  - Guthrie Robert Packer Hospital /ID# 261838, Sayre, Pennsylvania
  - TMA Headlands LLC /ID# 259800, Myrtle Beach, South Carolina
  - Carolina Endocrine Associates Llc /ID# 259640, North Charleston, South Carolina
  - Palmetto Clinical Research - Summerville /ID# 258845, Summerville, South Carolina
  - Chattanooga Medical Research /ID# 257631, Chattanooga, Tennessee
  - PMG Research of Knoxville /ID# 256854, Knoxville, Tennessee
  - University of Tennessee Health Science Center /ID# 259825, Memphis, Tennessee
  - Lifedoc Research /ID# 262975, Memphis, Tennessee
  - Mid State Endocrine Associates /ID# 259641, Nashville, Tennessee
  - Texas Diabetes and Endocrinology - Central Austin /ID# 255728, Austin, Texas
  - Texas Diabetes and Endocrinology - South Austin /ID# 255723, Austin, Texas
  - Brusco, Corpus Christi, TX /ID# 256746, Corpus Christi, Texas
  - North TX Endocrine Center /ID# 255737, Dallas, Texas
  - Research Institute Dallas /ID# 256126, Dallas, Texas
  - Academy of Diabetes, Thyroid and Endocrine /ID# 255735, El Paso, Texas
  - Diabetes and Thyroid Center of Ft. Worth /ID# 256781, Fort Worth, Texas
  - Juno Research /ID# 259238, Houston, Texas
  - Biopharma Informatic - Houston - Business Center Drive /ID# 256149, Houston, Texas
  - PlanIt Research, PLLC /ID# 259221, Houston, Texas
  - Endocrine and Psychiatry Cente /ID# 259631, Houston, Texas
  - Tekton Research - Irving /ID# 260988, Irving, Texas
  - Southern Endocrinology Associates /ID# 256795, Mesquite, Texas
  - Texas Diabetes and Endocrinology /ID# 255722, Round Rock, Texas
  - Northeast Clinical Research of San Antonio, LLC /ID# 256868, San Antonio, Texas
  - Diabetes & Glandular Disease Clinic /ID# 255734, San Antonio, Texas
  - Consano Clinical Research, LLC /ID# 256138, Shavano Park, Texas
  - Texas Valley Clinical Research /ID# 261476, Weslaco, Texas
  - Advanced Research Institute /ID# 259821, Ogden, Utah
  - The University of Vermont Medical Center /ID# 256533, South Burlington, Vermont
  - Virginia Endocrinology Research /ID# 259623, Chesapeake, Virginia
  - Richmond VA Medical Center /ID# 262386, Richmond, Virginia
  - Salem VA Medical Center /ID# 262387, Salem, Virginia
  - Rainier Clinical Research /ID# 255802, Renton, Washington
  - MultiCare Rockwood Clinic /ID# 255951, Spokane, Washington
  - MultiCare Institute for Research & Innovation /ID# 255954, Tacoma, Washington
- Puerto Rico (5):
  - Clinical Research Investigator Group, LLC /ID# 263177, Bayamón
  - ISIS Clinical Research Center /ID# 263182, Guaynabo
  - BRCR Global Puerto Rico /ID# 268231, San Juan
  - GCM Medical Group, PSC /ID# 263183, San Juan
  - Mindful Medical Research /ID# 263184, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-341